CLINICAL TRIAL: NCT07088211
Title: Sacituzumab Tirumotecan and Toripalimab in the First-line Treatment of Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma Patients With trop2 and CPS Positive: A Prospective, Single Arm, Phase II Trial
Brief Title: Sacituzumab Tirumotecan and Toripalimab in the First-line Treatment of HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, ren guoxin, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-T291
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Tirumotecan and Toripalimab (Experimental)
  Interventions: Drug: Sacituzumab Tirumotecan and Toripalimab

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan and Toripalimab — The dosing regimen for the combination of Sacituzumab Tirumotecan and Toripalimab is as follows: the recommended dose of Sacituzumab Tirumotecan is 5mg/kg, administered intravenously every 2 weeks, and Toripalimab is administered intravenously (without prophylactic medication), with a fixed dose of 240mg, and 3mg/kg is used for subjects with baseline body weight<50kg. Each infusion lasts for 30 minutes (not less than 20 minutes, not more than 60 minutes), administered once every 2 weeks. The subjects will continue to receive combination therapy with Sacituzumab Tirumotecan and Toripalimab until the termination criteria are met.

SUMMARY:
This study is a single center, non controlled, prospective phase II clinical trial to evaluate the efficacy and safety of Sacituzumab Tirumotecan and Toripalimab in the first-line treatment of recurrent/metastatic head and neck squamous cell carcinoma patients with trop2 and CPS positive. The participants would receive Sacituzumab Tirumotecan and Toripalimab until termination criteria are met.

DETAILED DESCRIPTION:
Despite advances in diagnosis and treatment, more than 65% of patients with head and neck squamous cell carcinoma still experience recurrence, metastasis, or both. Patients with locally recurrent head and neck cancer who are ineligible for salvage surgery, radiotherapy, or their combination have a very poor prognosis, similar to that of patients with distant metastatic head and neck cancer (survival of 6-9 months without treatment). Due to the limitations of previous radiotherapy (especially dose and irradiation fields) and the constraints of normal tissue tolerance, which restrict the feasibility and success of re-irradiation, systemic therapy with active drugs (platinum agents, taxanes, antifolates, and cetuximab) has become the cornerstone of palliative therapy. The choice between single-agent therapy or combination therapy (two or three drugs) depends on the toxicity of these drugs, the patient's performance status, comorbidities, frailty, age, symptoms, and characteristics related to previous treatment (disease stage, specific drugs, combination regimens, response, and time to progression). The phase III EXTREME (Erbitux in First-Line Treatment of Recurrent or Metastatic Head and Neck Cancer) trial demonstrated that adding cetuximab to fluorouracil plus platinum (cisplatin or carboplatin) chemotherapy significantly improved overall survival (10.1 months vs. 7.4 months; hazard ratio for death, 0.80; 95% CI, 0.64-0.99; P=0.04), progression-free survival (5.6 months vs. 3.3 months), and overall response rate (36% vs. 20%) compared with chemotherapy alone, thus supporting chemotherapy plus cetuximab as the first-line standard treatment. Unfortunately, cetuximab requires weekly administration, which can cause infusion reactions and skin reactions, resulting in poor quality of life for patients.

The discovery that regulating the immune system can induce regression of solid tumors has transformed our understanding and treatment of cancer. In particular, the successful development of programmed death receptor 1 (PD-1) immune checkpoint inhibitors has significantly influenced the treatment of head and neck squamous cell carcinoma. In patients with recurrent or metastatic head and neck cancer who have received platinum-based therapy, the anti-PD-1 antibodies pembrolizumab and nivolumab have achieved durable responses and improved survival. Therefore, the U.S. Food and Drug Administration (FDA) approved these two drugs for second-line treatment of advanced head and neck squamous cell carcinoma in 2016 and pembrolizumab for first-line treatment of advanced head and neck squamous cell carcinoma in 2019.

The use of pembrolizumab in first-line treatment of advanced head and neck squamous cell carcinoma is mainly based on the success of the phase 3 KEYNOTE-048 study. In the KEYNOTE-048 study, 882 previously untreated patients with recurrent or metastatic head and neck squamous cell carcinoma were randomly assigned to receive pembrolizumab monotherapy, pembrolizumab plus chemotherapy (fluorouracil and platinum agents), or the standard treatment regimen of fluorouracil plus platinum agents plus cetuximab (the regimen in the EXTREME trial). In patients with tumors expressing PD-L1 (using a combined positive score cutoff of ≥20% or ≥1%), both pembrolizumab monotherapy and pembrolizumab plus chemotherapy improved the primary endpoint of overall survival compared with the EXTREME regimen (see Supplementary Appendix for details). Compared with the EXTREME regimen, pembrolizumab had a lower response rate but more durable responses and fewer associated toxic effects. In the overall population not selected based on PD-L1, pembrolizumab monotherapy did not improve survival compared with the EXTREME regimen, while pembrolizumab plus chemotherapy improved survival (13.0 months vs. 10.7 months; hazard ratio for death, 0.77; 95% CI, 0.63-0.93; P=0.003).

Currently, numerous ongoing clinical trials are combining targeted therapy and immunotherapy. The rationale for these combination therapies is that the two therapies integrate different immunological and tumor biological mechanisms to enhance anti-tumor activity; in addition, some evidence suggests that targeted therapy can enhance certain links in the "cancer-immune cycle" (such as tumor antigenicity, T cell priming/transport/infiltration, etc.) and synergistically enhance immunotherapy. TROP2 (trophoblast cell surface antigen 2), a transmembrane glycoprotein, plays an important role in tumor occurrence and development by regulating calcium signaling pathways, cyclin expression, and cell adhesion functions. Studies have shown that TROP2 is highly expressed in head and neck squamous cell carcinoma (HNSCC), and its abnormal elevation is significantly associated with the invasive phenotype of tumor cells, lymph node metastasis, and poor prognosis of patients. Compared with normal tissues, the expression level of TROP2 in head and neck cancer tissues can be several to dozens of times higher, making it a promising target for targeted therapy. The expression level of Trop2 in head and neck squamous cell carcinoma (HNSCC) is high, with a positive rate of up to 86%, and it is associated with poor prognosis in patients.

The TROPiCS-03 basket study is an ongoing, open-label, multi-cohort, phase 2 study evaluating the anti-tumor activity and safety of the TROP2 ADC drug Sacituzumab Govitecan (SG) in patients with advanced solid tumors, including head and neck squamous cell carcinoma (HNSCC). A total of 43 adult patients with histologically confirmed locally recurrent or metastatic HNSCC who had disease progression after platinum-based chemotherapy and anti-PD-(L)1 inhibitor therapy (combined or sequential) were enrolled. The median duration of SG treatment for all patients was 2.5 months (0.3-12.3 months), and the median number of treatment cycles was 4 (1-17 cycles). The investigator-assessed ORR was 16%, all of which were partial responses (PR); the median DoR was 4.2 months, and the 6-month DoR rate was 43%. In terms of other secondary endpoints, the median PFS was 4.1 months, with 6-month and 12-month PFS rates of 32% and 12%, respectively; the median OS was 9.0 months, with 6-month and 12-month OS rates of 75% and 28%, respectively. In terms of safety, all patients experienced treatment-emergent adverse events (TEAEs) of any grade, the most common being diarrhea, nausea, and neutropenia, each occurring in 20 patients (47%). Grade 3 or higher TEAEs occurred in 25 patients (58%), the most common being neutropenia (33%), anemia (9%), and leukopenia (9%), indicating potential efficacy and safety in advanced head and neck cancer.

Trop2 ADC drugs can target and deliver cytotoxic drugs (such as topoisomerase I inhibitors SN-38 or DXd) to induce tumor cell death and release tumor-associated antigens (TAAs) and damage-associated molecular patterns (DAMPs, such as ATP, HMGB1, calreticulin). The released DAMPs bind to pattern recognition receptors on the surface of dendritic cells (DCs), promoting DC maturation and migration to lymph nodes, presenting tumor antigens to CD8⁺ T cells, and initiating adaptive immune responses. Therefore, there is a mechanism for combining Trop2 ADC drugs with PD-1 immunotherapy. Lukangsazumab is a TROP2-targeted ADC drug, which consists of an anti-TROP2 monoclonal antibody, a linker, and a cytotoxic drug (topoisomerase I inhibitor). Its mechanism of action is that the recombinant anti-TROP2 humanized monoclonal antibody specifically recognizes the TROP2 antigen on the surface of tumor cells, is endocytosed by tumor cells, and releases the payload intracellularly, inducing DNA damage in tumor cells, thereby leading to cell cycle arrest and apoptosis. In addition, the drug has a bystander effect, which can kill adjacent tumor cells and further enhance the anti-tumor effect. The OptiTROP-Lung01 study is a non-randomized controlled, phase II study evaluating the efficacy and safety of Lukangsazumab combined with the PD-L1 inhibitor KL-A167 as first-line treatment for driver gene-negative locally advanced or metastatic non-small cell lung cancer (NSCLC). A total of 103 patients were enrolled, divided into cohorts 1A and 1B, who received Lukangsazumab 5 mg/kg once every three weeks (Q3W) + KL-A167 1200 mg Q3W (cohort 1A) or Lukangsazumab 5 mg/kg once every two weeks (Q2W) + KL-A167 900 mg Q2W (cohort 1B) until disease progression or intolerable toxicity. The primary endpoint of the study was investigator-assessed ORR, and secondary endpoints included disease control rate (DCR), DoR, PFS, OS, and safety. As of the data cutoff date (January 2, 2024), the median follow-up time for cohort 1A and cohort 1B was 14.0 months and 6.9 months, respectively. Efficacy analysis results showed that the ORR of the Lukangsazumab + KL-A167 combination therapy regimen in cohort 1A (Q3W regimen) was 48.6% (18/37, with 16 confirmed responses), the median DoR was not reached, the DCR was 94.6%, the median PFS was 15.4 months (95% CI 6.7-NE), and the 6-month PFS rate was 69.2%. The ORR of the combination regimen in cohort 1B (Q2W regimen) was as high as 77.6% (45/58, with 40 confirmed responses), the DCR reached 100%, and both the median DoR and median PFS were not reached, with a 6-month PFS rate of 84.6%. These results demonstrate the potential value of PD-1 combined with TROP2 ADC drug therapy.

Toripalimab is an innovative biological product independently developed by Junshi Biosciences with complete independent intellectual property rights, and it is the first domestic PD-1 monoclonal antibody to receive conditional approval from the National Medical Products Administration (NMPA). Clinical trial results of toripalimab in various cancers such as malignant melanoma, nasopharyngeal carcinoma, and esophageal squamous cell carcinoma have shown that immune-related adverse events are rare. It received the first global conditional approval in China on December 17, 2018, for the treatment of unresectable or metastatic melanoma that was previously ineligible for systemic therapy. In head and neck squamous cell carcinoma, toripalimab combined with cetuximab is recommended in the 2024 CSCO guidelines for second-line or salvage treatment of recurrent metastatic head and neck squamous cell carcinoma.

Sacituzumab Tirumotecan is an independently developed drug by Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. It uses a proprietary Kthiol (pyrimidine-thiol) linker, which irreversibly conjugates with the anti-TROP2 monoclonal antibody at the antibody end and binds to a belotecan-derived topoisomerase I inhibitor at the toxin end, with a mean drug-to-antibody ratio (DAR) of up to 7.4. Based on its unique design, the payload of Sacituzumab Tirumotecan can be released through pH-sensitive cleavage in the tumor microenvironment or enzymatic hydrolysis in tumor cells, and it also has a bystander effect. High affinity, high targeting, triple anti-tumor effects, and appropriate stability ensure an effective balance between efficacy and safety. The TROPiCS-03 basket study enrolled 43 patients with histologically confirmed locally recurrent or metastatic HNSCC who had disease progression after platinum-based chemotherapy and anti-PD-(L)1 inhibitor therapy (combined or sequential). The investigator-assessed ORR was 16%, the median DoR was 4.2 months, and the 6-month DoR rate was 43%. In terms of safety, all patients experienced treatment-emergent adverse events (TEAEs) of any grade, the most common being diarrhea, nausea, and neutropenia, each occurring in 20 patients (47%). Grade 3 or higher TEAEs occurred in 25 patients (58%), the most common being neutropenia (33%), anemia (9%), and leukopenia (9%). Based on the data from this study, the dose of Sacituzumab Tirumotecan in head and neck cancer is 5 mg/kg.

Therefore, it is proposed to conduct a single-arm, phase II clinical study aimed at evaluating the safety and efficacy of Sacituzumab Tirumotecan combined with toripalimab as first-line treatment in patients with TROP2-positive, CPS ≥ 1 recurrent/metastatic head and neck squamous cell carcinoma, thereby providing a new treatment option for this patient population with extremely poor prognosis and no standard treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, regardless of gender; Histologically or cytologically confirmed newly diagnosed locally advanced, recurrent or metastatic head and neck squamous cell carcinoma (primary tumor sites include oropharynx, oral cavity, hypopharynx, and larynx) that cannot be cured by local treatment. No anti-tumor systemic treatment has been received in the recurrent or metastatic stage (systemic treatment as part of local advanced tumor treatment is allowed, provided that more than 6 months have passed from the end of treatment to the signing of informed consent); ECOG performance status of 0 or 1; Expected survival period ≥ 12 weeks; At least one measurable lesion according to RECIST 1.1 criteria. Lesions that have received previous radiotherapy can be used as measurable lesions if disease progression occurs; Availability of tumor tissue for PD-L1 detection (paraffin-embedded specimens within 2 years or fresh tumor tissue); PD-L1 CPS ≥ 1 and positive trop2 expression, detected by immunohistochemistry; For oropharyngeal cancer patients, P16 detection status, detected by IHC;

Normal function of major organs within 2 weeks before treatment, meeting the following criteria:

Bone marrow function: Hemoglobin ≥ 100g/L, white blood cell count ≥ 4.0×10^9/L or neutrophil count ≥ 2.0×10^9/L, platelet count ≥ 100×10^9/L without blood transfusion or colony-stimulating factor support; Liver function: Serum total bilirubin level ≤ 1.5 times the upper limit of normal, aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 times the upper limit of normal; Renal function: Serum creatinine level < 1.5 times the upper limit of normal or creatinine clearance rate ≥ 60ml/min, blood urea nitrogen ≤ 200mg/L; Urinary protein < +; if urinary protein is +, the 24-hour total protein must be < 500mg; Blood glucose: Within the normal range and/or for diabetic patients, blood glucose is controlled in a stable state during treatment; Cardiac function: No myocardial infarction within 1 year; no unstable angina; no symptomatic severe arrhythmia; no cardiac insufficiency; For women of childbearing age, serum pregnancy test results must be negative within 7 days before the first administration of the trial drug; males with reproductive capacity or females with the possibility of pregnancy must use highly effective contraceptive methods (such as oral contraceptives, intrauterine devices, abstinence, or barrier contraception combined with spermicides) throughout the trial, and continue contraception for 12 months after the end of treatment; Subjects voluntarily participate in this study, sign the informed consent form, have good compliance, and cooperate with follow-up; Patients whom doctors believe can benefit from the treatment.

Exclusion Criteria:

* Disease progression occurring within 6 months after systemic treatment for locally advanced head and neck squamous cell carcinoma; A history of primary nasopharyngeal carcinoma; Central nervous system metastasis and/or carcinomatous meningitis; Patients with hearing loss ≥ grade 2 or neuropathy ≥ grade 2 who are currently receiving anti-tumor treatment; Patients who have participated in or are participating in other drug/therapy clinical trials within 4 weeks before the first administration of the study drug; Patients who have received hematopoietic stimulating factors (such as granulocyte colony-stimulating factor (G-CSF), erythropoietin, etc.) within 1 week before the first administration of the study drug; Positive results for HIV antibody or Treponema pallidum antibody tests;

Patients with active hepatitis B or hepatitis C:

For those with positive HBsAg or HBcAb, additional HBV DNA testing is required (if the result is higher than the upper limit of the normal range); For those with positive HCV antibody test results, additional HCV RNA testing is required (if the result is higher than the upper limit of the normal range); Active lung diseases (interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or a history of active pulmonary tuberculosis; Patients with any active autoimmune disease or a history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; vitiligo that does not require systemic treatment can be included; asthma that has been completely relieved in childhood and requires no intervention in adulthood can be included; asthma in patients requiring medical intervention with bronchodilators cannot be included); Patients who are using immunosuppressants or systemic hormone therapy for the purpose of immunosuppression (dose > 10mg/day prednisone or other hormones with equivalent efficacy) and continue to use them within 2 weeks before enrollment;

Having any uncontrollable clinical problems, including but not limited to:

Persistent or active (severe) infections; Poorly controlled diabetes; Cardiac diseases (New York Heart Association class III/IV congestive heart failure or heart block); The following conditions occurring within 6 months before the first dose: deep vein thrombosis or pulmonary embolism; myocardial infarction; severe or unstable arrhythmia or angina pectoris; percutaneous coronary intervention, acute coronary syndrome, coronary artery bypass grafting; cerebrovascular accident, transient ischemic attack, cerebral embolism.

Large amounts of pleural effusion or ascites with clinical symptoms requiring symptomatic treatment; Patients who received cytochrome P450 3A4 (CYP3A4) inhibitors within one week before screening; A history of stem cell transplantation or organ transplantation; Patients with a history of psychoactive substance abuse who are unable to abstain or a history of mental disorders; Other severe, acute or chronic medical diseases or laboratory test abnormalities that the researcher judges may increase the risks related to study participation or may interfere with the interpretation of study results; Patients judged by the researcher to have poor compliance, or other conditions that make them unsuitable for participating in this trial; A history of other malignant tumors within 5 years, except for cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, early-stage prostate cancer, and carcinoma in situ of the cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 12 months
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.

SECONDARY OUTCOMES:
Progression Free Survival | 12 months
  PFS was defined as the time from enrollment to the first documented PD per RECIST 1.1, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD
overall survival | 12 months
  OS was defined as the time from enrollment to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Number of Participants Experiencing an Adverse Event (AE) | 12 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for each treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Yue He, M.D., Principal Investigator — the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China